CLINICAL TRIAL: NCT04306588
Title: Accessing Mobility Quality Using Wearable Sensors
Brief Title: Accessing Mobility Using Wearable Sensors
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The PI moved to another institution
Sponsor: Baylor College of Medicine (Other)
Collaborators: Michael E. DeBakey VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Bijan Najafi, PhD, Professor of Surgery, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 40765
Record Dates: First submitted 2020-03-09; First posted 2020-03-13 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: COPD; Pulmonary Disease; Pulmonary Restrictive Disease; Congestive Heart Failure; Cardiovascular Diseases
Keywords: COPD; CHF; Cardiovascular Diseases
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases; Heart Failure; Cardiovascular Diseases | interventions — Exercise; Telerehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tele-rehabilitation exercise Group (Experimental): Participants who are suffering from a chronic illness such as COPD or CHF and are referred for tele-rehabilitation intervention at the VA-Houston will be qualified for the purpose of this study.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Participants are undergoing a 12 weeks tele-rehabilitation program.
  Other Names: Tele-rehabilitation

SUMMARY:
This study will examine whether wearable sensors can be used to track changes in cognitive-motor performance in response to a disease or an intervention.

The investigators specific aims are twofold, first aim to explore whether and how a clinical condition such as Chronic obstructive pulmonary disease (COPD) or Congestive Heart Failure (CHF) may impact motor-cognitive performance measurable using validated wearable devices (e.g., LEGSys, BalanSENS, and Frailty Meter). Second, the investigators will explore whether an exercise intervention provided via tele-medicine (tele-rehabilitation) can enhance motor-cognitive performance.

DETAILED DESCRIPTION:
The investigators specific research questions: (1) Which motor-cognitive parameters measurable by wearable sensors (e.g. gait, balance, frailty index, etc) are linked to specific diseases (e.g. COPD, CHF) (2) Which motor-cognitive parameters are most responsive to identify changes in patients ambulatory performance related to Tele-rehabilitation

The investigators will recruit a minimum of 15 per clinical condition with a maximum of 150 per clinical condition in subjects suffering from different disorders, which may impact motor-cognitive. Targeted disorders: COPD and CHF. Other chronic illness may also be recruited such as Diabetes, Peripheral Arterial Disease, Morbus Parkinson, Cancer, Neuropathy, Frailty, Mild Cognitive Impairment, Depression, and patients undergoing major surgical intervention. Fifteen or more people with the same disorder would form a group.

The investigators will measure motor-cognitive performance from each subject. For this purpose several sensors will be attached to the body using elastic straps. Each subject will be asked to dedicate approximately 1 hour of their time for each visit. A series of health related questionnaires will be used to evaluate the quality of life, clinical problems, cognition, and pain intensity levels, respectively. Medical history (from the subject's chart) and demographic information will be obtained.

This study consists of Core and Ancillary Measurements. Core Measurements (Motor cognitive test) will be performed during all visits whereas Ancillary Measurements may not be required for anyone.

If the subject is undergoing tele-rehabilitation intervention, which may also benefit functional status (e.g. improvement in balance), the investigators will re-examine motor-cognitive performance using the test described above to evaluate the sensitivity of the proposed test in tracking outcomes in response to the intervention or predict outcomes based on baseline assessments. Specifically, depending on the type of intervention and frequency of standard of care visits for follow-up at the clinic, the investigators may re-assess functional performance at each follow-up standard of care visit, upon the availability of the subject. Please note that the number of follow up visits will not exceed 12 visits over the course of 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Any individual 18 years old or 65+ older is eligible to participate.
* Must be diagnosed with a chronic illness such as COPD or CHF.
* Should be refereed to one of the tele-rehabilitation program offered at VA-Houston.

The investigators will be enrolling veteran subjects

Exclusion Criteria:

* Non-ambulatory (unable to walk with or without assistance a distance of at least 10 meter).
* Unlikely to fully comply with the protocol (e.g., long-distance travel if multiple follow-up visits are required)
* Unwilling to provide informed consent.
* Severe visual and hearing problems who may not be able to interact with tele-rehabilitation.
* Unstable medical region (those who may change medication over next 12 weeks).
* Severe cognitive impairment and psychiatric problems who may not be able to follow tele-rehabilitation instructions based on judgement of clinical investigators.
* Participating in another active intervention that may affect cognitive-motor performance, and those who do not have capacity to consent.

The investigators will not exclude patients with internal devices such as a deep brain stimulator or electronic devices for pain management, but the investigators will not be placing Bioharness device in people with such conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-05-21 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline gait speed at 12 weeks | Baseline and 3 months
  Gait change from Baseline to 12 weeks
  The investigators will quantify gait speed using a validated wearable device, called LEGSys
Change from baseline balance at 12 weeks | Baseline and 3 months
  Balance will be quantified by measuring body sway during still upright standing for duration of 30 seconds. The investigators will use a validated wearable device, called BALANSens to measure body sway.
Change from baseline frailty index at 12 weeks | Baseline and 3 months
  Physical frailty is quantified by frailty index. Frailty index will be measured using a validated wearable device, called Frailty meter. scale is 0 to 1, higher value indicates more severity in frailty.

SECONDARY OUTCOMES:
Change from baseline Fear of Falling at 12 weeks | Baseline and 3 months
  Fear of falling is assessed using Fall Efficacy Scale International (FES-I) questionnaire. Scores range from 16 (no concern about falling) to maximum 64 (severe concern about falling).
Change from baseline depression at 12 weeks | Baseline and 3 months
  Depression will be assessed using Center of Epidemiologic Depression Scale (CES-D) questionnaire. Scores range from 0 to 60, with high scores indicating greater depressive symptoms. The CES-D also provides cutoff scores (e.g., 16 or greater) that aid in identifying individuals at risk for clinical depression.
Change from baseline cognitive performance at 12 weeks | Baseline to 3 months
  Cognitive performance will be assessed using Montreal Cognitive Assessment (MoCA). Scores on the MoCA range from zero to 30, with a score of 26 and higher generally considered normal.
Change from baseline functional performance at 12 weeks | Baseline to 3 months
  Functional Performance using 6 minute walk distance (6MWD) test
Change from baseline Risk of falling at 12 weeks | Baseline and 3 months
  Risk of falling will be assessed using timed Up and Go test
Change from baseline motor capacity at 12 weeks | Baseline and 3 months
  Motor capacity will be assessed by 5 times sit to stand test

CONTACTS AND LOCATIONS:
Overall Officials: Bijan Najafi, PhD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Michael E. DeBakey Veterans Affairs Medical Center, Houston, Texas, United States